CLINICAL TRIAL: NCT01396226
Title: A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled Phase II Study to Assess the Effects on Atrial and Ventricular Refractoriness of an Intravenous Infusion of AZD2927 in Patients Undergoing an Invasive Electrophysiological Procedure
Brief Title: A Multi-centre Study Comparing the Effects of AZD2927 and Placebo on the Electrical Activity in the Heart in Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: D4120C00002; 2011-001716-59 (EudraCT Number)
Record Dates: First submitted 2011-07-13; First posted 2011-07-18 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Arrhythmia
Keywords: Atrial refractoriness; cardiac electrophysiology; IKACh
MeSH Terms: conditions — Arrhythmias, Cardiac | interventions — AZD2927

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): A single dose of AZD2927 administered as an iv infusion
  Interventions: Drug: AZD2927
- 2 (Placebo Comparator): A single dose of placebo administered as an iv infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD2927 — A single dose of AZD2927 administered as an iv infusion
  Arms: 1
Drug: Placebo — A single dose of placebo administered as an iv infusion
  Arms: 2

SUMMARY:
Medical Products Agency

DETAILED DESCRIPTION:
* A Multi-Centre, Double-Blind, Randomised, Placebo-Controlled Phase II Study to Assess the Effects on Atrial and Ventricular Refractoriness of an Intravenous Infusion of AZD2927 in Patients Undergoing an Invasive Electrophysiological Procedure.
* The study has an adaptive design. In the 1st dose group the planned number of randomised patients is 24. The tentative number of randomised patients in the optional 2nd dose group is 12, 24 or 36 and thus a total maximum of 60 patients will be randomised in the study.

ELIGIBILITY:
Inclusion Criteria:

* male or postmenopausal female, aged 20 to 80 years inclusive,
* clinical indication for catheter ablation of atrial flutter,
* history of paroxysmal atrial flutter, with or without paroxysmal AF. Single episodes of persistent atrial flutter or AF requiring cardioversion do not exclude the patient from the study,
* sinus rhythm at randomisation,
* adequate anticoagulation or antithrombotic treatment according to ESC guidelines 2010 or national guideline,

Exclusion Criteria:

* cardioversion within 14 days before randomisation,
* history of stroke or transient ischaemic attack (TIA). History of significant head trauma, epilepsy or other disorders increasing the risk for seizures,
* QTcF >450 ms or <350 ms measured in sinus rhythm at randomisation,
* history and/or signs of clinically significant sinus node dysfunction. Sinus bradycardia (50 beats per minute or less) at randomisation,
* personal or family history of Torsades de Pointes (TdP), any other polymorphic ventricular tachycardia, long QT syndrome, short QT syndrome, Brugada syndrome, or personal history of sustained (>30 s) monomorphic ventricular tachycardia.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan C Carlsson, MD, PHD, Study Director — AstraZeneca; Hakan Walfridsson, MD, PHD, Principal Investigator — University Hospital Linkoping Sweden
Locations (5):
- Research Site, Oslo, Norway
- Sweden (4):
  - Research Site, Linköping
  - Research Site, Örebro
  - Research Site, Stockholm
  - Research Site, Umeå

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study had enrolled 20 patients. A total of 18 patients were randomised of which 12 patients received AZD2927. All patients who received treatment completed the study.
Groups:
- AZD2927: AZD2927 solution for infusion
- PLACEBO: Placebo solution for infusion
Period: Overall Study
Arm/Group | AZD2927 | PLACEBO
Started | 12 | 6
Patients Who Received Treatment | 12 | 6
Patients Who Completed Treatment | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD2927 | PLACEBO | Total
Number analyzed (Participants) | 12 | 6 | 18
Age Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (7.7) | 63.8 (8.3) | 59.9 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 11 | 5 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Left Atrial Effective Refractory Period
Description: Change in LAERP from before IP infusion to 1st and 2nd assessments during IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: Full A analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: msec
Groups:
- Arm 1 - AZD2927: AZD2927 solution for intravenous (i.v.) infusion
- Arm 2 - PLACEBO: Placebo solution for intravenous (i.v.) infusion
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec
  1st Assessment | 2.5 (8.9) | 5 (23)
  2nd Assessment | 2.5 (9.7) | 10.8 (34.4)

2. Secondary Outcome: Ventricular Effective Refractory Period
Description: Change in VERP from before IP infusion to 1st and 2nd assessments during IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec | -0.8 (9) | 1.7 (7.5)

3. Secondary Outcome: Paced QT Interval
Description: Change in CS Paced QT interval (P600 MS) from before and after IP infusion during electrophysiological measurements
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec | -0.9 (8.7) | 6.3 (8.4)

4. Secondary Outcome: Atrio-ventricular Effective Refractory Period
Description: Change from observation before IP infusion to during 1st and 2nd LAERP Mean
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 8 | 6
msec
  During IP 1st LAERP Mean | -16.9 (18.1) | 1.7 (18.1)
  During IP 2nd LAERP Mean | -19.4 (17.6) | 3.2 (16.5)

5. Secondary Outcome: PA Interval
Description: Reflects intra-atrial conduction and is defined as the interval from the onset of the P wave in the surface ECG to the onset of atrial activation (A) in the His bundle electrogram. Change from observation before IP infusion to 30 min after IP start
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec | 1.7 (12) | 9.3 (15.4)

6. Secondary Outcome: AH Interval
Description: Change from observation before IP infusion to 30 mins after IP start. AH interval- the conduction time from the low right atrium at the inter-atrial septum through the AV node to the His bundle, ie, intra-nodal conduction time.
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec | 0 (14.2) | -2.2 (12.1)

7. Secondary Outcome: HV Interval
Description: Change from observation before IP infusion to 30 mins after IP start. HV interval - represents conduction time from the proximal His bundle to the ventricular myocardium, ie, infra-nodal conduction time.
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec | -3.5 (8.9) | 3.5 (4.9)

8. Secondary Outcome: PR Interval
Description: Interval from the onset of the P-wave to the start of the QRS complex. Change from observation before IP infusion to 6 to 8 hours and 20 to 24 hours after IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec
  06:00-08:00 | -5.1 (17.0) | 19.3 (17.9)
  20:00-24:00 | -8.0 (18.6) | 4.3 (21.4)

9. Secondary Outcome: QRS Duration
Description: Change from observation before IP infusion to 6 to 8 hours and 20 to 24 hours after IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec
  06:00-08:00 | -1.2 (6.1) | -0.3 (8.5)
  20:00-24:00 | -2.5 (9.6) | -2.5 (7.3)

10. Secondary Outcome: RR Interval
Description: Change from observation before IP infusion to 6 to 8 hours and 20 to 24 hours after IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: FAS
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 12 | 6
msec
  06:00-08:00 | 21.3 (170.4) | 57.2 (74.2)
  20:00-24:00 | -11.5 (202) | -8.3 (139.9)

11. Primary Outcome: Left Atrial Effective Refractory Period
Description: Change in LAERP from before IP infusion to 1st and 2nd assessments during IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: Per Protocol (PP)
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 11 | 6
msec
  1st Assessment | 2.7 (9.3) | 5 (23)
  2nd Assessment | 2.7 (10.1) | 10.8 (34.4)

12. Secondary Outcome: Ventricular Effective Refractory Period
Description: Change in VERP from before IP infusion to 1st and 2nd assessments during IP infusion
Time Frame: Baseline to last assessment during IP infusion
Population: PP
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 11 | 6
msec | -0.9 (9.4) | 1.7 (7.5)

13. Secondary Outcome: Paced QT Interval
Description: Change in CS Paced QT interval (P600 MS) from before and after IP infusion during electrophysiological measurements
Time Frame: Baseline to last assessment during IP infusion
Population: PP
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Arm 1 - AZD2927 | Arm 2 - PLACEBO
Number analyzed (Participants) | 11 | 6
msec | -1.0 (9.1) | 6.3 (8.4)

ADVERSE EVENTS:
Arm/Group | AZD2927 | PLACEBO
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 2/12 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD2927 (N=12) | PLACEBO (N=6)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
MEDICAL DEVICE COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days